CLINICAL TRIAL: NCT03953872
Title: Current Status of Antihypertensive Drug Treatment in Non-cardiac Surgical Population
Brief Title: Antihypertensives in Non-cardiac Surgical Population
Status: Completed | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: antihypertensives 2019
Record Dates: First submitted 2019-04-27; First posted 2019-05-17 (Actual); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Perioperative Antihypertensive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- ARB: Group of angiotensin receptor blockers(ARB) monotherapy users. A subject was considered as an ARB user when the total prescription days of ARB monotherapy was at least 30.
- combination of CCB and ARB: Group of calcium channel blockers(CCB) and angiotensin receptor blockers(ARB) combination users. A subject was considered as a CCB and ARB combination user when the total prescription days of CCB and ARB combination therapy was at least 30.
- CCB: Group of calcium channel blockers(CCB) monotherapy users. A subject was considered as a CCB user when the total prescription days of CCB monotherapy was at least 30.
- No treatment: Group of nonusers of antihypertensives. A subject was considered as a nonuser never received regular antihypertensive treatment or total prescription days of antihypertensives was less than 30.

SUMMARY:
A cohort of hypertension patients undergoing elective non-cardiac surgery was constructed to investigate current status of antihypertensive drug treatment in non-cardiac surgical population.

DETAILED DESCRIPTION:
Perioperative changes in blood pressure (BP) are associated with perioperative risks. However, there is little information regarding the current status of antihypertensive treatment in non-cardiac surgical population. A cohort of 351 hypertension patients aged between 18 to 85-year old undergoing elective non-cardiac surgery was constructed to investigate the application of antihypertensive drugs, systemic involvement, perioperative hemodynamics and internal environment to grasp the perioperative impact of different antihypertensive drugs, and to further provide a reference for the preoperative antihypertensive strategy of surgery patients.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective non-cardiac surgery with hypertension(i.e., with a systolic blood pressure(SBP) of >=140 mmHg and/or a diastolic blood pressure(DBP) of >=90 mmHg based on the Seventh Report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure) or self-reported use of antihypertensive medication

Exclusion Criteria:

* Patients under the age of 18 years old
* Patients more than 85 years old
* Patients suspected of intracranial hypertension

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing elective non-cardiac surgery in Renji hospital
Sampling Method: Non-Probability Sample
Enrollment: 351 (Actual)
Dates: Start 2018-11-23 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
perioperative blood press(BP) | from the moment on arrival to the operating room until the moment leaving PACU, assessed up to 240 minutes.
  baseline BP before the operation, when entering and exiting post-anesthesia care unit(PACU)

SECONDARY OUTCOMES:
pH, base excess, and concentration of HCO3- in blood gases | 5 minutes after extubating in PACU
  arterial blood gases detected by using the ABL800 (Radiometer Med Aps Ltd, Copenhagen, Denmark)
the incidence of hypotension in PACU | from the moment on arrival to PACU until 60 minutes after arriving or the moment leaving PACU, whichever came first, assessed up to 240 minutes.
  If there were more than two consecutive episodes of hypotension (which was defined as SBP less than 80% of baseline) a "rescue" intravenous bolus of 100 mg of phenylephrine was given.
the incidence of hypertension in PACU | from the moment on arrival to PACU until 60 minutes after arriving or the moment leaving PACU, whichever came first, assessed up to 240 minutes.
  the incidence of hypertension, which was defined as SBP greater than 120% of baseline
hospitalization days | from the date of admission until the date of discharge or date of death from any cause, whichever came first, assessed up to 100 days
  The duration of this single episode of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Jie Chen, M.S., Study Chair — Renji Hospital, School of Medicine, Shanghai Jiaotong University, China
Locations (1):
- Renji Hospital, Shanghai Jiao Tong University, School of Medicine, Shanghai, Shanghai Municipality, China